CLINICAL TRIAL: NCT03812224
Title: A Phase 3 Japanese Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Erenumab in Migraine Prevention
Brief Title: A Controlled Trial of Erenumab in Migraine Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170609
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erenumab (Experimental): Participants were to receive erenumab 70 mg once a month for 24 weeks during the double-blind treatment period followed by erenumab 70 mg once a month for 28 weeks during the open-label treatment period.
  Interventions: Drug: Erenumab
- Placebo (Placebo Comparator): Participants were to receive placebo to erenumab once a month for 24 weeks during the double-blind treatment period followed by erenumab 70 mg once a month for 28 weeks during the open-label treatment period.
  Interventions: Drug: Erenumab; Drug: Placebo

INTERVENTIONS:
Drug: Erenumab — Administered by subcutaneous injection once a month
  Other Names: AMG 334; Aimovig®
Drug: Placebo — Administered by subcutaneous injection once a month
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the efficacy and safety of erenumab for prevention of migraine in Japanese adults with episodic migraine (EM) and chronic migraine (CM).

DETAILED DESCRIPTION:
Migraine prevention is an area of a large unmet medical need, with existing therapies often having modest efficacy and poor tolerability. Calcitonin gene-related peptide (CGRP) receptor antagonism is a novel approach to migraine preventive therapy. Erenumab is a human monoclonal antibody against canonical CGRP receptor. The present study is a phase 3 trial intended to assess the efficacy and safety of erenumab for prevention of migraine in Japanese adults with episodic migraine (EM) and chronic migraine (CM).

The study consists of a screening period (up to 7 weeks, including a 4-week baseline period), a 24-week double-blind treatment period (DBTP), a 28-week open-label treatment period (OLTP), and an 8-week safety follow-up period (12 weeks after the last dose of investigational product).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any study specific activities/procedures.
* Japanese subjects greater than or equal to 20 to less than or equal to 65 years of age upon entry into screening.
* History of migraine (with or without aura) for greater than or equal to 12 months before screening according to the International Headache Society Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018) based on medical records and/or patient self-report
* Migraine frequency: Chronic Migraine (CM) or Episodic Migraine (EM) over the 3 months before screening based on the following criteria:

  1. CM is defined as greater than or equal to 15 headache days per month of which greater than or equal to 8 headache days on average across the 3 months meet criteria as migraine days
  2. EM is defined as less than 15 headache days per month of which at least 4 or more headache days on average across the 3 months meet criteria as migraine days

Exclusion Criteria:

* Subjects greater than 50 years of age at migraine onset.
* History of cluster headache or hemiplegic migraine headache.
* Unable to differentiate migraine from other headaches.
* Migraine with continuous pain, in which the subject does not experience any pain-free periods (of any duration) during the 1 month before the screening period.
* Malignancy, except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years.

Other exclusion criteria may apply

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (34):
- Japan (34):
  - Research Site, Matsuyama, Ehime
  - Research Site, Kasuga-shi, Fukuoka
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Kahoku-gun, Ishikawa-ken
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Osaka, Osaka
  - Research Site, Toyonaka-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Iruma-gun, Saitama
  - Research Site, Saitama-shi, Saitama
  - Research Site, Tokorozawa-shi, Saitama
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Shimotsuga-gun, Tochigi
  - Research Site, Chofu-shi, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Tottori-shi, Tottori
  - Research Site, Yonago-shi, Tottori
  - Research Site, Toyama, Toyama
  - Research Site, Hofu-shi, Yamaguchi
  - Research Site, Yamaguchi, Yamaguchi
  - Research Site, Kai-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either
  1. the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or
  2. clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Hirata K, Takeshima T, Sakai F, Imai N, Matsumori Y, Tatsuoka Y, Numachi Y, Yoshida R, Peng C, Mikol DD, Lima GPDS, Cheng S. Early onset of efficacy with erenumab for migraine prevention in Japanese patients: Analysis of two randomized, double-blind, placebo-controlled studies. Brain Behav. 2022 Mar;12(3):e2526. doi: 10.1002/brb3.2526. Epub 2022 Feb 24. PMID 35201674
- [Background] Hiramatsu K, Onizuka Y, Hasebe M, Yoshida R, Numachi Y. Novel Drug for Migraine Prophylaxis: Mode of Action, Efficacy and Safety of Erenumab. Shinryo to Shinyaku (Med Cons New-Remed) 2021:58(11):797-832
- [Background] Hirata K, Sakai F, Takeshima T, Imai N, Matsumori Y, Yoshida R, Numachi Y, Peng C, Mikol DD, Cheng S. Efficacy and safety of erenumab in Japanese migraine patients with prior preventive treatment failure or concomitant preventive treatment: subgroup analyses of a phase 3, randomized trial. J Headache Pain. 2021 Sep 18;22(1):110. doi: 10.1186/s10194-021-01313-8. PMID 34537006
- [Background] Takeshima T, Sakai F, Hirata K, Imai N, Matsumori Y, Yoshida R, Peng C, Cheng S, Mikol DD. Erenumab treatment for migraine prevention in Japanese patients: Efficacy and safety results from a Phase 3, randomized, double-blind, placebo-controlled study. Headache. 2021 Jun;61(6):927-935. doi: 10.1111/head.14138. Epub 2021 Jun 21. PMID 34153117
- [Background] Hirata K, Takeshima T, Sakai F, Numachi Y, Yoshida R, Koukakis R, Hasebe M, Yui D, da Silva Lima GP, Cheng S. Long-term efficacy and safety of erenumab in Japanese patients with episodic and chronic migraine: results from a 28-week open-label treatment period of a randomised trial. BMJ Open. 2023 Aug 18;13(8):e068616. doi: 10.1136/bmjopen-2022-068616. PMID 37597868
- [Background] Kitamura S, Takeshima T, Yui D, da Silva Lima GP, Koukakis R, Peng C, Yoshida R, Numachi Y, Hasebe M. Efficacy of Erenumab for Migraine Prevention in Japanese Patients with Episodic and Chronic Migraine: Results of a Post-Hoc Pooled Analysis. Neurol Ther. 2023 Dec;12(6):1993-2006. doi: 10.1007/s40120-023-00538-w. Epub 2023 Sep 12. PMID 37698837
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 41 centers in Japan. The study consisted of a 24-week double-blind treatment period (DBTP), a 28-week open-label treatment period (OLTP), followed by an 8-week safety follow-up (12 weeks after the last dose of investigational product).
Pre-assignment Details: Eligible participants were randomized 1:1 to erenumab 70 mg or placebo. Randomization was stratified by migraine type (episodic migraine [EM] / chronic migraine [CM]) and migraine preventive treatment status (ever used [prior and/or current] or never used).
Groups:
- Placebo QM: Participants randomized to receive placebo once a month (QM) for 24 weeks during the double-blind treatment period followed by erenumab 70 mg once a month for 28 weeks during the open-label treatment period.
- Erenumab 70 mg QM: Participants randomized to receive erenumab 70 mg once a month for 24 weeks during the double-blind treatment period followed by erenumab 70 mg once a month for 28 weeks during the open-label treatment period.
Period: Double-blind Treatment Period
Arm/Group | Placebo QM | Erenumab 70 mg QM
Started | 131 | 130
Completed | 127 | 127
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Decision by Sponsor | 0 | 1
Period: Open-label Treatment Period
Arm/Group | Placebo QM | Erenumab 70 mg QM
Started | 127 | 127
Completed | 125 | 124
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Decision by Sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QM | Erenumab 70 mg QM | Total
Number analyzed (Participants) | 131 | 130 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.3) | 44.2 (8.5) | 44.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 111 | 227
  Male | 15 | 19 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 131 | 130 | 261
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 131 | 130 | 261
Migraine Type [Count of Participants; unit: Participants] — Episodic migraine is characterized by migraine with fewer than 15 headache days per month.
  Chronic migraine is characterized by 15 or more headache days per month (where at least 8 of those days are migraine days).
  Participants
    Episodic migraine | 80 | 79 | 159
    Chronic migraine | 51 | 51 | 102
Prior Migraine Preventive Treatment Status [Count of Participants; unit: Participants]
  Ever used (including prior and/or current users) | 100 | 100 | 200
  Never used | 31 | 30 | 61
Monthly Migraine Days [Mean (Standard Deviation); unit: days / month] — A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura, lasting for ≥ 4 hours and meeting protocol-specified criteria. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline period.
  days / month | 11.84 (5.70) | 12.40 (5.99) | 12.12 (5.84)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days (MMD) Over Months 4, 5, and 6 of the Double-blind Treatment Period
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura, lasting for ≥ 4 hours, and meeting at least 1 of the following criteria:
  1. ≥ 2 of the following pain features:
     * unilateral
     * throbbing
     * moderate to severe
     * exacerbated with exercise/physical activity
  2. ≥ 1 of the following associated symptoms:
     * nausea
     * vomiting
     * photophobia and phonophobia
  The change from baseline in monthly migraine days was calculated as the average number of migraine days per month during the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment period minus the number of migraine days during the 4-week baseline period.
Time Frame: 4-week baseline period and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment period
Population: The efficacy analysis set included randomized participants who received at least 1 dose of investigational product and had at least 1 change from baseline measurement in MMD during the DBTP. Observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: migraine days / month
Groups:
- Placebo QM: Participants received placebo once a month for 24 weeks during the double-blind treatment period.
- Erenumab 70 mg QM: Participants received erenumab 70 mg once a month for 24 weeks during the double-blind treatment period.
Arm/Group | Placebo QM | Erenumab 70 mg QM
Number analyzed (Participants) | 128 | 129
migraine days / month | -1.98 [-2.72 to -1.24] | -3.60 [-4.36 to -2.85]
Statistical Analysis 1: Comparison: Placebo QM vs Erenumab 70 mg QM; The primary endpoint was analyzed using a generalized linear mixed model which includes treatment, visit, treatment-by-visit interaction, stratification factors of migraine type and prior migraine preventive treatment status, and baseline value as covariates and assumes a first-order auto regression covariance structure; Test type: Superiority; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.62, 95% CI [-2.52 to -0.73]

2. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Mean Monthly Migraine Days Over Months 4, 5, and 6 of the DBTP
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine with or without aura, lasting for ≥ 4 hours, and meeting at least 1 of the following criteria:
  1. ≥ 2 of the following pain features:
     * unilateral
     * throbbing
     * moderate to severe
     * exacerbated with exercise/physical activity
  2. ≥ 1 of the following associated symptoms:
     * nausea
     * vomiting
     * photophobia and phonophobia
Time Frame: 4-week baseline period and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment period
Population: Efficacy analysis set; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QM | Erenumab 70 mg QM
Number analyzed (Participants) | 131 | 130
percentage of participants | 16.8 | 31.5
Statistical Analysis 1: Comparison: Placebo QM vs Erenumab 70 mg QM; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test, stratified by stratification factors of migraine type and prior migraine preventive treatment status; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.29 to 4.23]

3. Secondary Outcome: Change From Baseline in Mean Monthly Acute Migraine-specific Medication Treatment Days Over Months 4, 5, and 6 of the DBTP
Description: An acute migraine-specific medication treatment day is any calendar day during which a participant took a migraine-specific medication (e.g., triptan or ergotamine).
  The change from baseline in monthly acute migraine-specific treatment days was calculated as the average number of migraine-specific treatment days per month during the last 3 months of the 24-week double-blind treatment period minus the number of migraine-specific treatment days during the 4-week baseline period.
Time Frame: 4-week baseline period and the last 3 months (months 4, 5, and 6) of the 24-week double-blind treatment period
Population: Efficacy analysis set; observed data
Measure: Least Squares Mean (95% Confidence Interval); unit: days / month
Arm/Group | Placebo QM | Erenumab 70 mg QM
Number analyzed (Participants) | 128 | 129
days / month | -1.10 [-1.74 to -0.46] | -2.57 [-3.21 to -1.93]
Statistical Analysis 1: Comparison: Placebo QM vs Erenumab 70 mg QM; Analysis utilizes a generalized linear mixed model which includes treatment, visit, treatment-by-visit interaction, stratification factors of migraine type (episodic migraine or chronic migraine) and prior migraine preventive treatment status (ever used or never used), and baseline value as covariates and assumes a first-order auto regression covariance structure; Test type: Superiority; p < 0.001, Generalized Linear Mixed Model; LS Mean Difference = -1.47, 95% CI [-2.24 to -0.71]

ADVERSE EVENTS:
Time Frame: DBTP: From first dose of study drug up to the first dose of open-label study drug (24 weeks) for participants who entered the OLTP, or up to 12 weeks after the last dose (up to 32 weeks) for participants who did not enter the OLTP. OLTP: From first dose of study drug in the OLTP up to 12 weeks after last dose (up to 36 weeks).
Groups:
- Double-blind Treatment Period: Placebo QM: Participants received placebo once a month for 24 weeks during the double-blind treatment period.
- Double-blind Treatment Period: Erenumab 70 mg QM: Participants received erenumab 70 mg once a month for 24 weeks during the double-blind treatment period.
- Open-label Treatment Period: Erenumab 70 mg QM: Participants received erenumab 70 mg once a month for 28 weeks during the open-label treatment period.
Arm/Group | Double-blind Treatment Period: Placebo QM | Double-blind Treatment Period: Erenumab 70 mg QM | Open-label Treatment Period: Erenumab 70 mg QM
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/130 | 0/254
Serious Adverse Events (participants affected / at risk) | 2/131 | 2/130 | 7/254
Other Adverse Events (participants affected / at risk) | 40/131 | 44/130 | 62/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Placebo QM (N=131) | Double-blind Treatment Period: Erenumab 70 mg QM (N=130) | Open-label Treatment Period: Erenumab 70 mg QM (N=254)
Appendicitis (Infections and infestations) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Period: Placebo QM (N=131) | Double-blind Treatment Period: Erenumab 70 mg QM (N=130) | Open-label Treatment Period: Erenumab 70 mg QM (N=254)
Constipation (Gastrointestinal disorders) | 2 | 6 | 13
Nasopharyngitis (Infections and infestations) | 37 | 35 | 49
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03812224/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT03812224/SAP_001.pdf